CLINICAL TRIAL: NCT06640803
Title: Increasing Access to Evidence-Based CHR-P Assessment and Treatment Via Stepped-Care in Community-based Settings
Brief Title: Sacramento Clinical High Risk for Psychosis Stepped-Care Program
Acronym: SCIP Step
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Sacramento County Behavioral Health Services (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1989082; H79SM086150 (Other Grant/Funding Number: SAMHSA)
Record Dates: First submitted 2024-10-04; First posted 2024-10-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Clinical High Risk for Psychosis; Ultra High Risk for Psychosis
Keywords: psychosis; stepped-care; psychosis screening; community-based care; dissemination and implementation
MeSH Terms: conditions — Psychotic Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: This is a dissemination and implementation trial in which the study team is training staff at nine local community mental health centers to implement a screening protocol and stepped-care intervention. These clinics will be providing treatment and the study group will be evaluating it. There is no control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Behavioral Case Management (Experimental): Once youths are identified with a clinical high risk for psychosis (CHRp) syndrome they will begin a 2-year, 6 step intervention. They will be assessed every 6 months. If youths continue to meet CHRp criteria they will move into the next step. If they no longer meet criteria they exit the study and resume standard care. If they develop psychosis or reach the end of the 2-year intervention they can move to EDAPT, a psychosis specialty clinic or work with personnel to find a more appropriate clinical service.
  Interventions: Behavioral: Stepped-Care including Cognitive Behavioral Case Management

INTERVENTIONS:
Behavioral: Stepped-Care including Cognitive Behavioral Case Management — Step 1:assessment and feedback, general engagement strategies, assessment of needs and social determinants of health, begin case management, goal setting. Step 2: TAU. Initiation of team-based care at community clinics and 'enhanced monitoring'. Step 3: atheoretically-based stress management skills (stress thermometer, coping skills and coping plans), problem solving strategies. Step 4: targeted intervention for CHRp. Initiation of formulation-based CBT modules, therapy consultation groups with the UC Davis team (UCD), regular meetings between clinic leadership and UCD. Participants may switch providers to increase level of early psychosis specialization. Step 5: add prescriber consultation groups with UCD. Step 6: assessment of trauma and family conflict then Family-Focused Therapy, Trauma-Focused Cognitive Behavioral Therapy, or CBT for CHR at UCD. Termination: At 24 months, referral to UCD coordinated specialty care clinic or other appropriate service for those still CHRp+.
  Other Names: Cognitive Behavioral Therapy for those at clinical high risk for psychosis; team-based stepped-care

SUMMARY:
This is a dissemination and implementation study that is evaluating a stepped-care intervention for identifying and treating youths at clinical high-risk for psychosis within multiple community mental health centers.

DETAILED DESCRIPTION:
The study aims to increase the capacity to identify and treat youths at clinical high-risk for psychosis (CHRp) across Sacramento, CA by disseminating and implementing in community mental health clinics (CMHCs) universal screening and a stepped-care, team-based intervention that includes training and ongoing support in a Cognitive Behavioral Therapy package called Cognitive Behavioral Case Management (CBCM). The study is being conducted in nine non-psychosis specialty CMHCs across 5 agencies, all of which treat young people with public insurance (Medi-Cal/Medicaid) or no insurance. All youths aged 12-25 will be screened when beginning care and those who screen positive and agree will be assessed by the only specialty early psychosis clinic in the county, at the University of California-Davis. Thus the study also aims to triage this limited resource of specialized early psychosis expertise. CHRp+ youth will then begin a 2 year stepped-care intervention at their CMHCs and can move to the early psychosis specialty clinic if they still meet CHRp criteria after 2 years or develop psychosis. The specialty early psychosis service provides ongoing support and consultation.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical High Risk for Psychosis Syndrome as assessed by the mini-SIPS
2. Aged between 12-25 years old
3. Receiving care in one of six identified community mental health clinics
4. Eligibility for Sacramento County Medicare
5. Ability to provide informed consent

Exclusion Criteria:

1. Intellectual disability (IQ<70)
2. Urgent clinical need for a higher level of care

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 223 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility: The number of youth at clinical high risk for psychosis enrolled in stepped care over the course of the intervention. | 2, 3, or 4 years depending on site
  1. Duration of enrollment in the stepped-care intervention for young people identified as at clinical high-risk for psychosis through their community health setting.
Acceptability: Proportion of enrolled youths who move into each step of stepped-care | 2, 3, or 4 years depending on site
  Number of youth enrolled in stepped care at each assessment time point (0-, 6-, 12-, 18-, 24-month).
Reach: Universal screening outcomes | 2, 3, or 4 years
  Number of youths who reach each stage of the screening pipeline including:
  1. Number of youths screened.
  2. Number of screened youths who score positive on the screening measure (Prodromal Questionnaire Brief).
Reach: Number of community clinicians trained in specialized stepped care | 2, 3, or 4 years
  1. The number of clinicians employed at targeted community mental health agencies who complete training in Cognitive Behavioral Case management (CBCM).
  2. The number of these CBCM trained clinicians who enroll in the trial.
Effectiveness: Number of youth who meet criteria for a clinical high risk for psychosis (CHRp) syndrome at each step of the intervention. | from enrollment to the end of treatment at 2 years
  Number of youth who meet CHRp criteria on the Abbreviated Clinical Structured Interview for DSM-5 Attenuated Psychosis Syndrome (mini SIPS) and reach each stage of the intervention (baseline, 6-, 12-, 18-, 24-months).

SECONDARY OUTCOMES:
Modified Colorado Symptom Index (MCSI) | Baseline, 6-, 12-, 18-, 24-months, or study exit (up to 24 months)
  Self-report omnibus measure of symptom severity across multiple domains.
Global Impression Scale | Baseline, 6-, 12-, 18-, 24-months, or study exit (up to 24 months)
  Single item self-assessment of overall life function.
Global Functioning: Social and Role Scales | Baseline, 6-, 12-, 18-, 24-months, or study exit (up to 24 months)
  Clinician rated scales assessing social and role functioning.
Life and Treatment satisfaction | Baseline, 6-, 12-, 18-, 24-months, or study exit (up to 24 months)
  Self-report likert scale questions that assess overall functioning, symptom severity, and satisfaction with various aspects of the trial treatment.
Barriers and Facilitators interviews | 6 months after enrollment and when their final treatment client completes treatment
  Qualitative interviews with study clinicians and site leadership to identify barriers and facilitators to implementation.
Barriers and Facilitators Survey | 6 months after clinician's enrollment and again when their final client completes care
  Survey created by study investigators to accompany qualitative interviews and assess opinions on the appropriateness and effectiveness of Cognitive Behavioral Case Management and stepped-care in this setting.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - River Oak Center for Children, Elk Grove, California
  - Turning Point Community Programs, Elk Grove, California
  - University of California Department of Psychiatry and Behavioral Sciences; Early Psychosis Programs, Sacramento, California
  - University of California-Davis CAARE Diagnostic and Treatment Center, Sacramento, California
  - Capital Star Community Services, Sacramento, California
  - Heartland Child and Family Services, Sacramento, California

IPD SHARING:
Plan to Share IPD: Undecided
Screening and treatment provided in this study occur at community mental health centers by community providers and is embedded within their care models. Sites are protective of data generated from the treatment consumers who are participating in this trial and each have asked to make their own determinations about data sharing.